CLINICAL TRIAL: NCT05386979
Title: Multimodal Analgesic Management of Naborphine Combined With Opioid Free Under General Anesthesia in OSA Patients Undergoing Weight Loss Surgery Under the Concept of ERAS: a Prospective, Randomized, Parallel Controlled Study
Brief Title: Multimodal Analgesic Management of Naborphine Combined With Opioid Free Anesthesia in OSA Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YXLL-KY-2022(035)
Record Dates: First submitted 2022-05-10; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Analgesics，Opioid; Bariatric Surgery
Keywords: Opioid free anesthesia; Bariatric Surgery; ERAS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid anesthesia group (Other): Anesthesia induction with propofol 2.5mg/kg, rocuronium bromide 0.6mg/kg, sufentanil 0.3μg/kg, intubation was performed when BIS value reached 40-60. Intraoperative pump injection of propofol 4-12 mg/kg·h and remifentanil 0.2-0.5 μg/kg·min to maintain anesthesia. Ultrasound-guided transversus abdominis plane block (with 0.375% ropivacaine 40ml) will be implemented preoperatively. Ondansetron 8mg and sufentanil 10 μg will be given after surgery. For PCA, sufentanil 2μg/kg + dexmedetomidine 2μg/kg + ondansetron 24mg.
  Interventions: Procedure: Opioid free anesthesia technology
- Opioid free anesthesia group (Experimental): Anesthesia induction with propofol 2.5mg/kg, rocuronium bromide 0.6mg/kg, naborphine 0.2mg/kg，esketamine 0.3mg/kg, intubation was performed when BIS value reached 40-60. Intraoperative pump injection of propofol 4-12 mg/kg·h and esketamine 0.3～0.5mg/kg·h. Ultrasound-guided transversus abdominis plane block (with 0.375% ropivacaine 40ml) will be implemented preoperatively. Ondansetron 8mg and naborphine 0.2mg/kg will be given after surgery. For PCA, naborphine 2mg/kg + dexmedetomidine 2μg/kg + ondansetron 24mg.
  Interventions: Procedure: Opioid free anesthesia technology

INTERVENTIONS:
Procedure: Opioid free anesthesia technology — We have adopted a variety of methods to replace the use of opioids in the process of balanced anesthesia.

SUMMARY:
Comparative study to explore the effect of opioid free anesthesia technology in perioperative analgesia management, clarify the effect of naborphine instead of opioids on perioperative analgesia management in morbid obesity patients with moderate and severe OSA, reduce related adverse events, and explore the latest clinical anesthetic drugs.

DETAILED DESCRIPTION:
1. The concept of enhanced recovery after surgery (ERAS) has been applied in the perioperative period of many operations. Reducing the dosage of opioids is an important part of the concept of ERAS.
2. Opioid free anesthesia technology has been recognized in reducing nausea and vomiting, but whether it can meet the perioperative analgesic needs of patients undergoing bariatric surgery and obtain more clinical benefits still has no research supportment.
3. This study is expected to clarify the clinical effect of opioid free anesthesia technology in perioperative analgesia management of morbid obesity patients with moderate and severe OSA, reduce adverse events, and explore the latest clinical anesthesia scheme.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade I ~ III;
2. Age from 18 - 65 years old;
3. BMI ≥ 35kg / m2 in patients with OSA to undergo bariatric surgery； （4 provide written informed consent for participation.

Exclusion Criteria:

1. Age < 18 years or age >65 years old;
2. Pregnancy test was positive;
3. Patients with a history of drug abuse or dependence on opioids;
4. Patients with chronic pain or severe heart, lung, liver or nervous system diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
postoperative NRS score | Score from the end of the operation and follow-up at the time point specified in the scoring form for a total of 27 hours.
  A subjective psychometric response scale used to measure distinct behavioral or physiological phenomena based on linear numerical gradient or yes/no alternatives. The Numeric Pain Scale (NRS) pain numerical score(0-10 score, 0: no pain, 10: worst imaginable pain). A pain measurement list about quiet NRS score and cough NRS score at different postoperative time will be used.

SECONDARY OUTCOMES:
Dosage of remedial analgesics postoperatively | It takes about 24 hours.
  If the participant still feels severe pain after operation and needs additional analgesic drugs for treatment, we will record the type and dose of drugs used by the patient.
Hemodynamic fluctuation | From the beginning of the general anesthesia induction to the time leaving PACU, it takes about 4 hours.
  Hemodynamic fluctuation during perioperative period. The levels of SBP in mmHg, DBP in mmHg, MAP in mmHg and HR in times/minute in basic(T0), after induction(T1), preoperative(T2) and after establishing pneumoperitoneum(T3) 1h after the pneumoperitoneum(T4) and Immediately after operation(T5), Before(T6) and after(T7) extubation were recorded.
Ramsay scale | Score from the end of the operation and follow-up at the time point specified in the scoring form for a total of 27 hours.
  Ramsay scale is the most widely used sedation scoring standard in clinic, which is simple and practical. This scale has multiple advantages: it is reproducible, easily executed and has good applicability. This has made the scale the most widely used to assess level of sedation for procedures in pediatrics. It is divided into six levels(1-6): 1 shows patient is anxious and agitated or restless, or both; 2 shows patient is co-operative, oriented, and tranquil; 3 shows patient responds to commands only; 4 shows patient exhibits brisk response to light tactile stimuli or loudauditory stimulus; 5 shows patient exhibits sluggish response to light tactile stimuli or loud auditory stimulus; 6 shows patient exhibits no response.
recovery time | It will take up to 1 hour or 2 hours.
  From the time when the patient entered PACU to the time when the participant meets the standard of leaving the PACU.
The levels of C-reactive protein (CRP) | It takes about 24 hours.
  We will collect the participant's blood at the time before surgery(T0), after surgery(T1), and 24h after surgery(T2) to obtain the levels of C-reactive protein (mg/L).
The levels of cortisol (COR). | It takes about 24 hours.
  We will collect the participant's blood at the time before surgery(T0), after surgery(T1), and 24h after surgery(T2) to obtain the levels of cortisol (nmol/L).
The levels of blood glucose (BG) | It takes about 24 hours.
  We will collect the participant's blood at the time before surgery(T0), after surgery(T1), and 24h after surgery(T2) to obtain the levels of blood glucose (mmol/L).
The levels of interleukin-6 (IL-6). | It takes about 24 hours.
  We will collect the participant's blood at the time before surgery(T0), after surgery(T1), and 24h after surgery(T2) to obtain the levels of IL-6 (pg/mL).
Scores of 15-item Quality of Recovery (QoR-15) scale 24 hours postoperatively of participants. | One day after the surgery.
  The QoR-15 scale is a validated tool to assess the quality of postoperative recovery (QoR) from 0 to 150. The QoR was classified as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) or poor (QoR-15 < 90).
Rate of postoperative nausea and vomiting | It takes about 24 hours.
  Postoperative nausea and vomiting will be recorded if it happens.
Acceptability of participants with laryngeal mask 24 hours after surgery. | One day after the surgery.
  One day after surgery, we will record the acceptability of laryngeal mask and the degree of postoperative pharyngeal pain of the participants. Acceptability of participants with laryngeal mask will be assessed by whether the participant was willing to receive laryngeal mask anesthesia again. Pharyngeal pain can be evaluated using the Numeric Pain Scale (NRS) pain numerical score. A subjective psychometric response scale used to measure distinct behavioral or physiological phenomena based on linear numerical gradient or yes/no alternatives. The Numeric Pain Scale (NRS) pain numerical score(0-10 score, 0: no pain, 10: worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Sun, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Yongtao Sun, Jinan, Shandong, China

REFERENCES:
- [Derived] Guo Y, Chen L, Gao Z, Zhang M, Liu M, Gao X, Liu Y, Zhang X, Guo N, Sun Y, Wang Y. Is esketamine-based opioid-free anesthesia more superior for postoperative analgesia in obstructive sleep apnea patients undergoing bariatric surgery? A study protocol. Front Med (Lausanne). 2022 Nov 15;9:1039042. doi: 10.3389/fmed.2022.1039042. eCollection 2022. PMID 36457567